CLINICAL TRIAL: NCT03394404
Title: ECG-I Phenotyping of Persistent AF Based on Driver Distribution to Predict Response to Pulmonary Vein Isolation
Acronym: PHENOTYPE-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 218367-1
Record Dates: First submitted 2017-12-04; First posted 2018-01-09 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation
Keywords: ECG-I Mapping Pulmonary Vein Isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ECG-I mapping and PVI (Experimental): ECG-I mapping and PVI
  Interventions: Device: ECG-I mapping and PVI

INTERVENTIONS:
Device: ECG-I mapping and PVI — ECG-I mapping and PVI

SUMMARY:
Atrial fibrillation (AF) is an irregular heart rhythm associated with significant morbidity and mortality. The pulmonary veins (the blood vessels carrying blood from the lungs into the left atrium) have been shown to send electrical signals into the heart that can cause and maintain AF. Pulmonary vein Isolation (PVI) is an established treatment where catheters are passed into the atria of the heart to deliver lines of scar to electrically isolate the pulmonary veins preventing them from transmitting these electrical signals into the left atrium.

The ECG-I is a system which involves wearing a jacket with many ECG electrodes to record electrical activity from the surface of the body. A CT scan then shows where these electrodes are relative to the atria, and computer modelling is used to reconstruct the movements of electricity on the surface of the heart and therefore identifying where the drivers (tissue causing and maintaining AF) are located.

Unfortunately, not all patients respond to PVI due to the drivers of AF being located in areas other than within the Pulmonary Veins. Identifying the drivers of AF is very difficult and the role they play has yet to be proved scientifically.

The investigators intend to enroll 100 patients with persistent AF and perform atrial mapping using the ECG-I system. Solely pulmonary vein isolation will be performed. Patients will be followed up to see if the distribution of drivers as predicted by the ECG-I predicts outcomes. This may improve patient selection for this procedure.

DETAILED DESCRIPTION:
Atrial Fibrillation (AF) is the commonest heart rhythm disturbance and is associated with significant morbidity and mortality. Catheter ablation (CA) is a procedure where catheters (leads) are passed into the heart and energy is used to disrupt and isolate (by freezing or cauterising) heart tissue causing AF. CA is an established therapy for AF. Success rates for CA for paroxysmal AF lies in the region of 70% or better. However, success rates for persistent AF is much lower and estimates lie in the region of 30-60%.

Current CA protocols for AF centre on isolating the pulmonary veins (the pulmonary veins drain into the left atrium) which have been proven to trigger AF. Pulmonary Vein Isolation (PVI) ablation alone seems sufficient to remove the trigger for the vast majority of patients with paroxysmal AF. However, in patients with persistent AF it is common for AF to continue after the pulmonary veins have been electrically isolated.

The difference in success rates between the paroxysmal and persistent form of AF is thought to be due to changes within the heart atria after AF has been established for some time. In persistent AF the atria dilate and remodel structurally and electrically, and therefore the maintenance of persistent AF differs from paroxysmal AF.

Persistent AF is thought to be maintained by focal sources, whether rotors or sites of radial activation. Currently, targeting other sites within the atria in addition to PVI such as fractionated electrograms (areas of electrical activity) are thought to be imprecise and require extensive ablation. Often AF will persist despite targeting additional sites within the atria.

One particular challenge is to select patients likely to benefit from CA. CA carries an approximate less than 1% risk of life threatening complication. Therefore being able to select suitable patients is desirable in order to prevent unnecessary procedures.

Currently clinical characteristics of patients or structural imaging have limited accuracy in selecting patients likely to benefit from CA. Mapping studies have shown that patients with persistent AF who have higher frequency signals near the pulmonary veins than being distributed in the left atrial body are more likely to terminate to sinus rhythm (normal heart rhythm) with PVI alone and to maintain sinus rhythm.

Studies have suggested that patients undergoing standard PVI ablation procedures for persistent AF who have coincidental interruption of drivers have a far better long term outcome. This suggests that the characteristics of atrial heart tissue and electrical activation patterns maintaining AF are likely to determine the response to ablation therefore it may be possible to determine more directly and accurately the likelihood of success by performing non-invasive mapping of the atria using the ECG-I.

It appears that a proportion of patients with persistent AF will maintain sinus rhythm long term after undergoing AF CA with standard PVI protocols alone. PVI can now be achieved quickly and safely using technologies such as the Cryoballoon (A freezing technology). Identification of patients that are likely to respond to PVI alone is therefore of great interest as it (1) identifies patients that may respond to a conservative strategy, and (2) in the absence of an effective strategy beyond PVI may allow de-selection of patients unlikely to benefit from ablation at all.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Persistent AF (i.e. episodes of AF that are continuous for > 1 week or have required DC cardioversion)
2. Willing for ablation.
3. Age between 18 to 80.
4. left atrial diameter <5 cm
5. left ventricular function >40%.
6. New York Heart Association class < 3.

Exclusion Criteria:

* Persistent AF diagnosed > 2 years ago
* left atrial diameter > 5 cm
* Severe left ventricular impairment (EF < 40%)
* New York Heart Association class 3 or 4 heart failure
* Known hypertrophic cardiomyopathy, cardiac sarcoid, or arrythmogenic ventricular cardiomyopathy.
* Known inherited arrhythmia such as Brugada or long QT syndromes
* Valvular disease that is more than moderate
* History of valve replacement (metallic or tissue)
* History of congenital heart disease (other than patent foramen ovale)
* Previous left atrial ablation (percutaneous or surgical)
* Cardiac surgery or percutaneous coronary intervention within the last 3 months.
* Myocardial infarction or unstable angina within the last 3 months.
* Unwillingness for ablation
* Unwillingness to be involved in study
* Suspected reversible cause of AF
* Any other contraindication to catheter ablation
* Age < 18 yrs or > 80 years
* Pregnancy
* Morbid obesity (defined as BMI >40)
* Any other medical problem likely to cause death within the next 18 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Freedom from Atrial Arrhythmia and association with distribution of drivers of AF | Performed 12-14 months post procedure
  All patients will undergo mapping with ECG-I during their procedure. The number of drivers and their locations will be collected. Patients who remain free from AF at 12 months will be compared to patients who relapsed comparing the number and location of these drivers.

SECONDARY OUTCOMES:
Impact of pulmonary vein isolation on drivers of AF | During AF Catheter Ablation
  Patients will undergo ECG-I mapping of their AF at baseline and then immediately after pulmonary vein isolation. The number of drivers and locations will be collected at both points and these will be compared to assess the impact of PVI.

CONTACTS AND LOCATIONS:
Overall Officials: Ross Hunter, Principal Investigator — Barts Heart Centre
Locations (1):
- Barts Heart Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dhillon GS, Honarbakhsh S, Graham A, Abbass H, Welch S, Daw H, Sporton S, Providencia R, Chow A, Earley MJ, Lowe M, Lambiase PD, Schilling RJ, Hunter RJ. ECG-I phenotyping of persistent AF based on driver burden and distribution to predict response to pulmonary vein isolation (PHENOTYPE-AF). J Cardiovasc Electrophysiol. 2022 Nov;33(11):2263-2273. doi: 10.1111/jce.15644. Epub 2022 Aug 16. PMID 35924481
- [Derived] Dhillon GS, Ahluwalia N, Honarbakhsh S, Graham A, Creta A, Abbass H, Chow A, Earley MJ, Lambiase PD, Schilling RJ, Hunter RJ. Impact of adenosine on mechanisms sustaining persistent atrial fibrillation: Analysis of contact electrograms and non-invasive ECGI mapping data. PLoS One. 2021 Mar 25;16(3):e0248951. doi: 10.1371/journal.pone.0248951. eCollection 2021. PMID 33765054
- [Derived] Dhillon GS, Schilling RJ, Honarbakhsh S, Graham A, Abbass H, Waddingham P, Sawhney V, Creta A, Sporton S, Finlay M, Providencia R, Chow A, Earley MJ, Lowe M, Lambiase PD, Hunter RJ. Impact of pulmonary vein isolation on mechanisms sustaining persistent atrial fibrillation: Predicting the acute response. J Cardiovasc Electrophysiol. 2020 Apr;31(4):903-912. doi: 10.1111/jce.14392. Epub 2020 Mar 1. PMID 32048786